CLINICAL TRIAL: NCT03510559
Title: A Comparison of Forearm Versus Brachial Plexus Blockade for Routine Hand and Wrist Surgery
Brief Title: Forearm vs Brachial Plexus Blockade for Routine Hand and Wrist Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-6152-A
Record Dates: First submitted 2018-03-06; First posted 2018-04-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Post-operative Pain Management
MeSH Terms: interventions — Brachial Plexus Block

STUDY DESIGN:
Intervention Model Description: Patients scheduled for ambulatory hand surgery will be assessed in the pre-operative assessment clinic at the time of surgical booking for recruitment into the study by their surgeon. A research assistant will then speak with the patient regarding the study in order to obtain informed consent for their participation.
  If the patient consents to participate in the study, they will be randomized into either the brachial plexus or forearm nerve block groups. The research assistants will be blinded as to the patient's allocation and during block performance to minimize bias.
Who Masked: Outcomes Assessor
Masking Description: The research assistants who will be performing the follow-up assessments of the patient will be blinded as to block group allocation. No other members of the team will be blinded for this study due to methodological constraints as the end result of these blocks is very different due to upper arm weakness expected with brachial plexus blocks, but not with forearm blocks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachial Plexus Block (Active Comparator): It will be at the discretion of the anesthesiologist performing the block to choose a supraclavicular, infraclavicular or axillary block to achieve adequate surgical anesthesia of the operative arm. After sterile skin preparation with chlorhexidine, a linear array transducer probe is placed on the skin and the appropriate nerve structures are identified. Local anesthetics (30 mL of 50:50 mix of 0.5% bupivacaine and 2% lidocaine) will then be injected in 5 mL aliquots after negative aspiration for blood to achieve circumferential spread around the brachial plexus. Patients who have a failed brachial plexus block may undergo a rescue forearm block, and will be recorded as requiring supplemental local anesthetic.
  Interventions: Drug: Brachial Plexus Block
- Forearm Nerve Block (Experimental): Patients allocated to the forearm block will have it performed in the semi-setting position. After sterile skin preparation with chlorhexidine and infiltration with 1 mL of 1% lidocaine, a linear array transducer probe is placed at the distal forearm to visualize each peripheral nerve (radial, ulnar, median, and lateral antebrachial cutaneous). A 5 cm 22 G insulated needle is then used to target each nerve individually and infiltrate 7.5mL of the 50:50 mixture (similar to the brachial plexus block group) at each nerve to a total of 30mL.
  Interventions: Drug: Forearm Nerve Block

INTERVENTIONS:
Drug: Forearm Nerve Block — Blockade of the arm below the elbow using local anesthetic (0.5% bupivacaine and 2% lidocaine) deposited under ultrasound guidance to facilitate performance of the surgical procedure.
  Arms: Forearm Nerve Block
Drug: Brachial Plexus Block — Blockade of the entire arm using local anesthetic (0.5% bupivacaine and 2% lidocaine) deposited under ultrasound guidance to facilitate performance of the surgical procedure.
  Other Names: Bracial Plexus Nerve Block
  Arms: Brachial Plexus Block

SUMMARY:
It is very common to perform nerve blocks for hand and wrist surgery. It allows the surgeon to perform the surgery and helps with pain control after surgery. This also means only light sedation is needed for the procedure instead of a general anesthetic, which speeds up recovery time.

There are 2 types of nerve blocks that can be done for hand and/or wrist surgery. The one that is done commonly now is where the whole arm is frozen with local anesthetic. Another option is to have a nerve block where only the arm from the elbow down is frozen. Either of these types of nerve blocks can be chosen to safely accomplish surgery of the hand or wrist. However, the best nerve block for hand and/or wrist surgery has not been decided yet.

In order to determine which block is best, the investigators will be looking at patient satisfaction with the experience, as well as the surgical conditions provided and overall safety.

It is thought that many patients may prefer the arm block below the elbow as it allows for greater mobility immediately following surgery, and the surgical conditions provided will be very similar to those of the full arm nerve block.

DETAILED DESCRIPTION:
A randomized controlled trial involving adult patients undergoing surgery to the wrist and hand with centralized random allocation of patients to 2 groups: 1)Brachial plexus block and 2)Forearm block. The brachial plexus group will undergo a standard brachial plexus block. The forearm group will undergo a block of the proximal forearm targeting the radial sensory, ulnar, median and lateral antebrachial cutaneous nerves.

Group allocation will not be blinded from the treating physicians or patients due to methodological constraints. However, the research assistants performing follow-up assessments will be blinded.

Brachial plexus anesthesia provides a reliable sensorimotor block for upper extremity surgery. It is the current gold standard of anesthesia for surgery on the hand. A forearm block is an alternative anesthetic technique. As day surgery for hand procedures is less invasive and has fewer analgesic requirements, it may be that a forearm block, which allows for preservation of upper extremity function, is of benefit for these types of procedures. It is anticipated that patients may appreciate the forearm block as opposed to a brachial plexus block as they will have greater functionality post-operatively upon returning home. This contrasts with a brachial plexus block which causes a flaccid and insensate upper extremity lasting for many hours beyond the surgical procedure longer than the anticipated analgesic requirements which may be detrimental. Conversely, a forearm block may not provide sufficient anesthesia to create a dense motor blockade, which may result in unwanted intra-operative hand movements during surgery. This could pose a significant safety concern.

A forearm block has successfully been used as a primary anesthetic in patients undergoing hand surgery, although no information has been published about patient satisfaction and events related to patient safety.

The investigators aim to assess patient satisfaction, as well as overall efficacy and safety of the forearm blocks for hand and wrist surgery, as compared to the gold standard of brachial plexus blocks.

ELIGIBILITY:
Inclusion Criteria:

* Consented, English-speaking, adult patients (age > 18)
* American Society of Anesthesiologists (ASA) classification I-III
* BMI ≤ 38 kg/m2 (quality of US imaging deteriorates significantly with obesity)
* Patients undergoing hand and/or wrist surgery (except wrist arthroscopy)

Exclusion Criteria:

* Previous upper extremity nerve block
* Contra-indication to nerve blocks e.g., infection, bleeding diathesis, allergy to local anesthetics
* Existing chronic pain disorders or history of use of ≥ 30mg morphine or equivalent per day
* Pre-existing neurological deficits or peripheral neuropathy involving the operative upper extremity
* Pregnancy
* Any significant psychiatric conditions that may affect patient assessment
* Inability to tolerate a forearm tourniquet
* Wrist arthroscopy surgery (requires upper arm tourniquet)
* Inability to speak or understand English without an interpreter present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with overall block | Study coordinators will assess QoR-15 change between baseline and 24 hours after surgery
  The impact of surgical and anesthetic interventions on perioperative quality of life will be assessed using the QoR-15 tool (Quality of Recovery -15). The QoR-15 is a patient-based outcome measure in the form of a 15-item validated questionnaire.

SECONDARY OUTCOMES:
Amount of intraoperative sedation required | 6 hours
  Intraoperative sedation required by the surgical time in minutes ( from operation room arrival to discharge) for varying surgical durations
Supplemental local anesthetic to block | 2 hours
  Requirement for additional local anesthetic in the block room from the block room arrival to discharge
Supplemental local anesthetic to block in operation room | 6 hours
  Requirement for additional local anesthetic intraoperatively (mL) from operation room arrival to discharge
Time in PACU | 6 hours
  Time spent in the post-operative anesthetic care unit measured in minutes from moment of PACU arrival to discharge
Surgical procedure time (minutes) | 6 hours
  Time spent completing the surgical procedure measured in minutes from time of incision until time of surgical dressing application
Block procedure time (minutes) | 2 hours
  Time spent completing the nerve block measured in minutes from time of initial ultrasound probe contact with skin until removal of needle at block completion
Analgesia provided by the nerve block | 6 hours
  Postoperative pain severity at rest will be assessed using a numerical rating scale (NRS; 0=no pain, 10=worst pain imaginable) score during the post-anesthesia care unit (PACU) stay.
Analgesia provided by the nerve block | 24 hours
  Postoperative pain severity at rest will be assessed using a numerical rating scale (NRS; 0=no pain, 10=worst pain imaginable) score at 24 hours post-op. Cumulative oral analgesic consumption since hospital discharge will also be measured at this time
Number and severity of safety-events as measured by hand movements recorded intraoperatively | 24 hours
  Assessing number and severity of intraoperative hand movements from time of incision until time of surgical dressing application

CONTACTS AND LOCATIONS:
Overall Officials: Ahtsham Niazi, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No